CLINICAL TRIAL: NCT06831617
Title: AI-based Low Dose CBCT Reconstruction for Lung Puncture Guidance: A Multicenter Randomized Controlled Study
Brief Title: AI-based Low Dose CBCT Reconstruction for Clinical Application
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AI guidance-Lung 001
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Lung Nodule
Keywords: Artificial Intelligence; Lung Nodule; Cone Beam CT; Lung Puncture; Images Reconstruction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI based CBCT reconstructed images guided lung puncture (Experimental): Participants in the experimental group undergo AI-based low dose (radiation dose is 1/6th of the dose used in the clinic) CBCT reconstructed images guided lung puncture procedures.
  Interventions: Other: AI-based low dose CBCT reconstructed images system
- Conventional CBCT images guided lung puncture (Placebo Comparator): Participants in the experimental group undergo conventional CBCT images guided lung puncture procedures.
  Interventions: Other: Conventional CBCT images system

INTERVENTIONS:
Other: AI-based low dose CBCT reconstructed images system — Participants in the experimental group undergo AI-based low dose (radiation dose is 1/6th of the dose used in the clinic) CBCT reconstructed images guided lung puncture procedures.
  Arms: AI based CBCT reconstructed images guided lung puncture
Other: Conventional CBCT images system — Participants in the experimental group undergo conventional CBCT images guided lung puncture procedures.
  Arms: Conventional CBCT images guided lung puncture

SUMMARY:
The goal of this clinical trial is to learn if AI-based low dose CBCT reconstructed images can guide lung puncture effectively. The main questions it aims to answer are:

1. Does the AI-based low dose CBCT reconstruction model reconstruct high quality images?
2. Is it possible that low-dose CBCT reconstructed images can guide lung puncture procedures without compromising the efficiency of the procedure? Researchers will compare AI-based low dose CBCT reconstructed images to a placebo (conventional CBCT images) to see if AI-based low dose CBCT reconstructed image can guide lung puncture procedures without compromising the efficiency of the procedure.

Participants will:

1. Undergo lung puncture under AI-based low dose CBCT reconstructed images guidance or under conventional CBCT images
2. Be followed up for 1 week postoperative to obtain patient complications

ELIGIBILITY:
Inclusion Criteria:

* Participants who require CBCT-guided precutaneous lung puncture (PLP) and meet the clinical indications for the procedure.
* Participants whose physical condition is suitable for PLP.
* Participants are willing to sign informed consent.

Exclusion Criteria:

* Participants have metallic implants in the body, which severely affects the image quality.
* Participants are pregnant or breastfeeding.
* Participants are unwilling or unable to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of puncture needles of participants undergoing percutaneous lung puncture procedures. | From enrollment to the end of the lung puncture procedure.
  The number of punctures was defined as the number of punctures performed throughout the percutaneous lung puncture procedure.

SECONDARY OUTCOMES:
Radiation Dose | From enrollment to the end of the lung puncture procedure.
  Radiation dose was defined as the radiation dose generated throughout the percutaneous lung puncture procedure.
Intraoperative and postoperative complications of participants undergoing lung puncture procedures | From enrollment to the end of the lung puncture procedure at 1 week.
  Intraoperative and postoperative complications were defined as those arising in parricipants during percutaneous lung puncture and within 7 days after puncture.

OTHER OUTCOMES:
Algorithmic performance (peak signal-to-noise ratio) | Through study completion, an average of 9 months.
  Peak signal-to-noise ratio (PSNR) is a metric used to measure the quality of an image or video, assessing the degree of distortion by comparing the peak signal power to the mean square error (MSE) between the original signal and the compressed or processed signal. PSNR is measured in decibels (dB), with higher values indicating less distortion and better image or video quality.
Algorithmic performance (structural similarity) | Through study completion, an average of 9 months.
  Structural similarity (SSIM) is a metric for evaluating the similarity of two images. SSIM value is between 0 and 1, the larger the value, the more similar the images are.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Wuhan Union Hospital, Wuhan, Hubei
  - Wuhan Union Jinyinhu Hospital, Wuhan, Hubei
  - Wuhan Union West Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No
The anonymized data is available from Huangxuan Zhao upon reasonable request.

REFERENCES:
- [Result] Zhao H, Xu Z, Chen L, Wu L, Cui Z, Ma J, Sun T, Lei Y, Wang N, Hu H, Tan Y, Lu W, Yang W, Liao K, Teng G, Liang X, Li Y, Feng C, Nie T, Han X, Xiang D, Majoie CBLM, van Zwam WH, van der Lugt A, van der Sluijs PM, van Walsum T, Feng Y, Liu G, Huang Y, Liu W, Kan X, Su R, Zhang W, Wang X, Zheng C. Large-scale pretrained frame generative model enables real-time low-dose DSA imaging: An AI system development and multi-center validation study. Med. 2025 Jan 10;6(1):100497. doi: 10.1016/j.medj.2024.07.025. Epub 2024 Aug 19. PMID 39163857